CLINICAL TRIAL: NCT01355289
Title: A Phase II, Randomized, Multicenter, Placebo-Controlled, Double-Blind, Parallel-Group Study, With an Open-Label Extension, to Evaluate the Efficacy, Safety, and Pharmacokinetics of E5501 in Subjects With Chronic Hepatitis C Virus Related Thrombocytopenia Who Are Potential Candidates for Antiviral Treatment
Brief Title: Chronic Hepatitis C Virus Related Thrombocytopenia to Evaluate the Effects of E5501
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E5501-G000-203
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Thrombocytopenia
Keywords: Chronic Hepatitis C related
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag; telaprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Core Study) (Placebo Comparator): Placebo, will be administered orally, once daily for up to 21 days.
  Interventions: Drug: Placebo
- Avatrombopag 10 mg (Core Study) (Active Comparator): Avatrombopag 10 mg, will be administered orally, once daily, preferably with food for up to 21 days.
  Interventions: Drug: Avatrombopag
- Avatrombopag 20 mg (Core Study) (Active Comparator): Avatrombopag 20 mg, will be administered orally, once daily, preferably with food for up to 21 days.
  Interventions: Drug: Avatrombopag; Drug: Pegylated interferon (PEG-IFN); Drug: Telaprevir; Drug: Ribavirin
- Avatrombopag 30 mg (Core Study) (Active Comparator): Avatrombopag 30 mg, will be administered orally, once daily, preferably with food for up to 21 days.
  Interventions: Drug: Avatrombopag
- Avatrombopag (Open-Label Extension) (Experimental): Avatrombopag will be initiated at a dose of 20 mg, once daily in the open-label extension (OLE) period. The avatrombopag dose will be titrated up or down in accordance with the participant's individual response, within the range of a minimum of 5 mg and a maximum of 50 mg for up to 48 weeks.
  Interventions: Drug: Avatrombopag; Drug: Pegylated interferon (PEG-IFN); Drug: Telaprevir; Drug: Ribavirin

INTERVENTIONS:
Drug: Avatrombopag
  Other Names: E5501; Avatrombopag maleate
  Arms: Avatrombopag (Open-Label Extension); Avatrombopag 10 mg (Core Study); Avatrombopag 20 mg (Core Study); Avatrombopag 30 mg (Core Study)
Drug: Placebo
  Arms: Placebo (Core Study)
Drug: Pegylated interferon (PEG-IFN) — Participants in Treatment Periods A2, B2, and B3 are to receive antiviral treatment PEG-IFN, ribavirin, or telaprevir. Provided by the sponsor.
  Arms: Avatrombopag (Open-Label Extension); Avatrombopag 20 mg (Core Study)
Drug: Telaprevir — Participants in Treatment Periods A2, B2, and B3 are to receive antiviral treatment PEG-IFN, ribavirin, or telaprevir. Provided by the sponsor
  Other Names: Incivek; Incivo
  Arms: Avatrombopag (Open-Label Extension); Avatrombopag 20 mg (Core Study)
Drug: Ribavirin — Participants in Treatment Periods A2, B2, and B3 are to receive antiviral treatment PEG-IFN, ribavirin, or telaprevir. Provided by the sponsor
  Other Names: Virazole; Rebetol; Copegus; Ribasphere; Moderiba dose pack; Moderiba
  Arms: Avatrombopag (Open-Label Extension); Avatrombopag 20 mg (Core Study)

SUMMARY:
To evaluate the efficacy of E5501 by measuring platelet response in subjects with chronic hepatitis C virus (HCV)-related thrombocytopenia who require antiviral treatment.

DETAILED DESCRIPTION:
This study had three phases: Prerandomization (Screening), Randomization (Core Study), and Open-Label Extension (OLE). The Randomization Phase included Treatment Periods A1 and A2 and a Follow-up Period (for those participants not continuing into the OLE phase). The OLE Phase included Treatment Periods B1, B2, and B3 (depending on when a participant entered the OLE), and a Follow-up Period. Participants may have been followed for sustained viral response, if appropriate. In the Core Study (randomization phase) participants were randomized (in a 1:1:1:1 ratio) to receive one of four treatments (placebo or avatrombopag [10mg, 20mg, and 30mg] for up to 21 days. Participants who successfully completed Treatment Period A1, (platelet count >=100x10^9/L) initiated antiviral treatment with pegylated interferon (PEG-IFN) alpha-2a and progressed to Treatment Period A2. Participants with a platelet count >=150x10^9/L initiated antiviral treatment and progressed into Treatment Period B2, study drug was interrupted then eventually restarted at 10 mg daily once their platelet counts returned to acceptable levels. Those who were not considered successful after 21 days in Treatment Phase A1 were withdrawn from the Core Study (Part A) and were eligible to enter the OLE at Treatment Period B1. Participants who chose to not enter the OLE entered into the Follow-up Phase. At the end of Treatment Period A2, eligible participants could enter the OLE at Treatment Period B3. In the OLE Phase, participants entering into Open-label Treatment Period B1 began once-daily treatment with avatrombopag at a dose of 20 mg without titration for up to 21 days. Once the participant's platelet counts were sufficient, they entered Treatment Period B2. Participant's eligible to enter into Treatment Period B2 received avatrombopag and antiviral treatment for 13 weeks. Participants who successfully completed Treatment Period A2 or B2 could continue on antiviral treatment for up to a maximum of 48 weeks (including the 13 weeks in Treatment Periods A2 or B2) and open-label avatrombopag, at the investigator's discretion. In Treatment Period B3, the dose of avatrombopag was allowed to be titrated up or down in accordance with the participant's platelet count response, within the range of a minimum of 5 mg and a maximum of 50 mg. In the Follow-up Period, participants were seen at either a single 30-day follow-up visit or followed for the full 30 days after the last dose of avatrombopag.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females greater than or equal to 18 years of age
2. Women of childbearing potential must agree to use a highly effective method of contraception for at least one menstrual cycle prior to starting study drug, throughout the entire study period, and for 30 days after the last dose of study drug
3. Subjects with chronic HCV-related thrombocytopenia (defined as a platelet count greater than or equal to 20x10^9/L to 70x10^9/L) who require antiviral treatment
4. Chronic HCV infection (defined as the presence of anti-HCV antibodies and detectable serum HCV RNA levels)
5. Model for End-stage Liver disease score greater than or equal to 24
6. Adequate renal function as evidenced by a calculated creatinine clearance greater than or equal to 50 mL/minute per the Cockcroft and Gault formula
7. Life expectancy greater than or equal to 3 months

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Any history of arterial or venous thrombosis, including partial or complete thrombosis (e.g., stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), thrombosis (partial or complete) in the main portal vein and portal vein branches, and thrombosis of any part of the splenic-mesenteric system
2. Any evidence of current portal vein thrombosis (PVT) as detected by Doppler sonography and portal vein flow rate less than 15 cm/second at Screening or within 30 days prior to Screening (revised per Amendment 02)
3. Any known family history of hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency)
4. Evidence of myocardial infarction in the last 6 months or uncompensated congestive heart failure (New York Heart Association Class III or IV)
5. Co-infection with human immunodeficiency virus (HIV) or hepatitis B or acute hepatitis C
6. Any prohibited concomitant medications or therapy that cannot be discontinued by Visit 1, e.g., subjects currently receiving interferon who cannot undergo a 4-week washout period prior to Screening, or subjects who receive blood products that affect platelet count within 1 week prior to Screening (revised per Amendment 02)
7. Weekly alcohol intake greater than 21 units (168 g) [male] and greater than 14 units (112 g) [female]
8. Any known medical condition, other than chronic liver disease, that can lead to thrombocytopenia
9. History of hepatocellular carcinoma, metastatic liver cancer, or liver transplantation (revised per Amendment 01) (revised per Amendment 02)
10. History of idiopathic thrombocytopenic Purpura (ITP)
11. History of myelodysplastic syndrome
12. History of pernicious anemia or subjects with vitamin B12 deficiency (defined as less than the lower limit of normal [LLN]) who have not had pernicious anemia excluded as a cause (Added per Amendment 02)
13. Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that, in the opinion of the investigator, could affect the subject's safety or study conduct
14. Subjects with a history of suicide attempts
15. Subjects with a history of hospitalization for depression within the past 5 years
16. Subjects with any current severe or poorly controlled psychiatric or seizure disorder
17. Current use of recreational drugs
18. Subjects who have participated in another investigational study within 30 days prior to Visit 1
19. Subjects with hypersensitivity, intolerance, or allergy to E5501 or any anti-HCV therapies or their ingredients
20. Any past or current (revised per Amendment 01) medical condition that, in the opinion of the investigator, would compromise the subject's ability to safely complete the study
21. Scheduled for surgery during the projected course of the study
22. Subjects who have any medical conditions or diseases that would contraindicate treatment with anti-HCV therapy (added per Amendment 01)
23. Subjects who are currently treated with proton pump inhibitors (PPIs) or H2-antagonist therapy but have not been receiving a stable dose for at least 6 weeks prior to randomization or have not completed these therapies more than 2 weeks prior to randomization (added per Amendment 01)
24. Fasting gastrin-17 blood levels exceeding 1.5 times the upper limit of normal (ULN) at Screening (including subjects on PPIs or H2 antagonists) (revised per Amendment 02)
25. Subjects with a history of gastric atrophy (added per Amendment 02)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Manhuchehri, Study Director — Eisai Inc.
Locations (2):
- United States (2):
  - Health Care Consultants, Los Angeles, California
  - Metropolitan Research, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Screening Period encompassed 14 days ±7 days. Prerandomization assessments took place in all participants who had provided informed consent.
Groups:
- Placebo (Core Study): Placebo, was given orally for up to 21 days once daily.
- Avatrombopag 10 mg (Core Study): Avatrombopag 10 mg, was administered orally, once daily, preferably with food for up to 21 days.
- Avatrombopag 20 mg (Core Study): Avatrombopag 20 mg, was administered orally, once daily, preferably with food for up to 21 days.
- Avatrombopag 30 mg (Core Study): Avatrombopag 30 mg, was administered orally, once daily, preferably with food for up to 21 days.
- Avatrombopag (Open Label Extension): Avatrombopag was initiated at a dose of 20 mg, once daily in the open label extension (OLE) period. The avatrombopag dose was titrated up or down in accordance with their individual response within the range of a minimum of 5 mg and a maximum of 50 mg for up to 48 weeks.
Period: Core Study
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study) | Avatrombopag (Open Label Extension)
Started | 17 | 16 | 18 | 14 | 0
Completed | 16 | 16 | 18 | 12 | 0
Not Completed | 1 | 0 | 0 | 2 | 0
Not completed — Adverse Event, Non-Fatal | 1 | 0 | 0 | 0 | 0
Not completed — Inadequate Therapeutic Effect | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0
Period: Open Label Extension
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study) | Avatrombopag (Open Label Extension)
Started | 0 | 0 | 0 | 0 | 62
Completed | 0 | 0 | 0 | 0 | 28
Not Completed | 0 | 0 | 0 | 0 | 34
Not completed — Adverse Event, Non-Fatal | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Inadequate Therapeutic Effect | 0 | 0 | 0 | 0 | 29
Not completed — Other | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Core Study): Placebo, was given orally for upto 21 days once daily.
- Total: Total of all reporting groups
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study) | Total
Number analyzed (Participants) | 17 | 16 | 18 | 14 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (7.96) | 55.3 (8.06) | 54.9 (7.38) | 53.6 (7.26) | 53.5 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants] — Full analysis set (FAS), the group of all randomized participants of core study.
  Participants
    Female | 3 | 4 | 5 | 5 | 17
    Male | 14 | 12 | 13 | 9 | 48

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline of Local Platelet Count by Visit During Treatment Period A1 of Core Study
Description: Missing platelet counts were imputed using last observation carried forward (LOCF) approach for subjects who achieved platelet response at prior visits.
Time Frame: Day 7 and Day 14
Population: Full analysis set (FAS), the group of all randomized participants of core study.
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study)
Number analyzed (Participants) | 17 | 16 | 18 | 14
cells x 10^9/L
  Day 7 | -0.1 (7.15) | 19.8 (17.59) | 26.5 (22.06) | 30.9 (37.65)
  Day 14 | -0.2 (13.79) | 29.2 (18.32) | 57.2 (31.39) | 55.4 (37.47)

2. Secondary Outcome: Number of Participants Who Achieved Platelet Count Greater Than 30 X 10^9/L From Baseline to Day 21 During Treatment Period A1 of Core Study
Description: Blood draws were taken to monitor platelet counts.
Time Frame: Baseline to Day 21
Population: Full analysis set (FAS), the group of all randomized participants of core study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study)
Number analyzed (Participants) | 17 | 16 | 18 | 14
Participants
  Yes | 1 | 9 | 16 | 11
  No | 16 | 7 | 2 | 3

3. Primary Outcome: Number of Participants Who Achieved Platelet Response (Greater Than or Equal to 100 x 10^9/L) by Day 21 of Treatment Period A1 of Core Study
Description: A responder was defined as a participant having a platelet count of greater than or equal to 100x10^9/L by Day 21 starting from an average baseline platelet count of greater than 20 x 10^9/L to less than or equal to 70 x 10^9/L.
Time Frame: Baseline to Day 21
Population: Full analysis set (FAS), the group of all randomized participants of core study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study)
Number analyzed (Participants) | 17 | 16 | 18 | 14
Participants
  Yes | 1 | 6 | 12 | 9
  No | 16 | 10 | 6 | 5
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Avatrombopag 10 mg (Core Study); Test type: Superiority or Other; p = 0.0236, Cochran-Mantel-Haenszel; Difference in % of Responders = 31.62, 95% CI 2-sided [5.39 to 57.84]
Statistical Analysis 2: Comparison: Placebo (Core Study) vs Avatrombopag 20 mg (Core Study); Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; Difference in % of Responders = 60.78, 95% CI 2-sided [36.30 to 85.27]
Statistical Analysis 3: Comparison: Placebo (Core Study) vs Avatrombopag 30 mg (Core Study); Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; Difference in % of Responders = 58.4, 95% CI 2-sided [30.92 to 85.88]

4. Secondary Outcome: Number of Participants Who Initiated Antiviral Treatment by Day 21 of Period A1 of Core Study
Description: Blood draws were taken to monitor platelet counts during the first 21 days of study treatment. When a platelet count of greater than or equal to 100 X 10^9/L was attained, antiviral treatment was initiated.
Time Frame: Baseline to Day 21
Population: Full analysis set (FAS), the group of all randomized participants of core study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study)
Number analyzed (Participants) | 17 | 16 | 18 | 14
Participants
  Yes | 1 | 6 | 13 | 9
  No | 16 | 10 | 5 | 5

ADVERSE EVENTS:
Time Frame: For each participant, treatment emergent adverse events were collected from the first day of administration of study drug up to 30 days after the last dose of study drug or up to approximately 2.5 years.
Description: Core Study Safety Analysis Set (SAS): All participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. OLE Safety Analysis Set: All participants who received at least 1 dose of avatrombopag study drug (either in the Core Study or the Extension Phase) and had a postdose safety assessment.
Arm/Group | Placebo (Core Study) | Avatrombopag 10 mg (Core Study) | Avatrombopag 20 mg (Core Study) | Avatrombopag 30 mg (Core Study) | Avatrombopag (Open Label Extension)
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/16 | 0/18 | 1/14 | 13/64
Other Adverse Events (participants affected / at risk) | 6/17 | 11/16 | 12/18 | 11/14 | 55/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Core Study) (N=17) | Avatrombopag 10 mg (Core Study) (N=16) | Avatrombopag 20 mg (Core Study) (N=18) | Avatrombopag 30 mg (Core Study) (N=14) | Avatrombopag (Open Label Extension) (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Core Study) (N=17) | Avatrombopag 10 mg (Core Study) (N=16) | Avatrombopag 20 mg (Core Study) (N=18) | Avatrombopag 30 mg (Core Study) (N=14) | Avatrombopag (Open Label Extension) (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 21
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 14
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 2 | 20
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6
Abdominal Pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 4 | 2 | 20
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 8
Asthenia (General disorders) | 0 | 1 | 2 | 1 | 8
Chills (General disorders) | 1 | 3 | 3 | 1 | 13
Fatigue (General disorders) | 0 | 1 | 3 | 2 | 16
Influenza like illness (General disorders) | 2 | 1 | 4 | 3 | 11
Injection site erythema (General disorders) | 0 | 1 | 1 | 0 | 6
Irritability (General disorders) | 0 | 0 | 1 | 1 | 7
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 6
Pyrexia (General disorders) | 1 | 0 | 2 | 2 | 9
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 4
Headache (Nervous system disorders) | 1 | 0 | 3 | 2 | 12
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 5
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 2 | 15
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 12
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Congenital lymphoedema (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Liver tenderness (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0
Food aversion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other